CLINICAL TRIAL: NCT04771325
Title: Assessment of the Effectiveness of Continuous Labour Support by a Trained Companion of Choice on Events of Labor and Maternal Satisfaction in the Bugisu Sub Region, Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: Swedish International Development Cooperation Agency (SIDA) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-54
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Labor Long
Keywords: Support, companion,labour

STUDY DESIGN:
Intervention Model Description: Educational; training of lay persons on support during labour
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Other): Women are normally escorted to the health facilities by one or more family members and or friends. Women usually labor in an open first stage room where more than one woman is admitted sometimes with curtains to separate the beds with one person allowed besides her to provide support. The support persons do not have designated roles to play during this process. Routine analgesia is not given neither is continuous fetal monitoring. Midwives,
  Interventions: Behavioral: Support from a trained companion
- Arm 2 (Experimental): One session of training on admission in labor. The training will focus on emotional and physical support; emotional support including being Present, demonstrating a caring and positive attitude, saying calming verbal expressions, using humor, praise, encouraging and acknowledging efforts during the process of pushing the baby. Physical support including supporting her to change position favoring upright positions, walking with her, giving her drinks and food, massage, reminding her to go and pass urine, helping her find a comfortable position for pushing, wipe her face with cool cloth and help her breast feed
  Interventions: Behavioral: Support from a trained companion

INTERVENTIONS:
Behavioral: Support from a trained companion — Birth companions trained on how to effectively support women during labor

SUMMARY:
A randomized control trial employing a cross sectional stepped wedge design. Women with anticipated vaginal delivery, receiving usual care for the control group while women receiving usual care plus support from a trained companion will constitute the experimental group. Events and outcomes will then be assessed during and after birth.

DETAILED DESCRIPTION:
The order of introduction of the intervention will be determined randomly. Control data will be obtained from the first health facility until the sample size for the control for that facility is achieved. Following collection of control data for the first facility, the intervention will be introduced to the same facility to a new group of participants. Simultaneously control data from the other facilities will be collected and this will be done until all the facilities are covered in a step wedge manner.

The intervention will consist of a session of training on admission in labor. The training will focus on emotional and physical support; emotional support including being Present, demonstrating a caring and positive attitude, saying calming verbal expressions, using humor, praise, encouraging and acknowledging efforts during the process of pushing the baby. Physical support including supporting her to change position favoring upright positions, walking with her, giving her drinks and food, massage, reminding her to go and pass urine, helping her find a comfortable position for pushing, wipe her face with cool cloth and help her breast feed.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a singleton fetus and a supposed cephalic presentation.
2. Women with a female friend or relative willing to stay with them through the process of labor and birth.

Exclusion Criteria:

* Women with a multiple pregnancy.
* Women with a previous cesarean section
* Women who are mentally incapacitated or deaf and dumb

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 535 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of a Spontaneous Vaginal delivery | labour duration
  delivery of the baby naturally without use of oxytocin, vacuum extraction, or a cesarean section

SECONDARY OUTCOMES:
coping and anxiety | labour duration
  Women's self-reported anxiety on admission and after birth will be measured using the 10 cm Visual Analogue Scales Coping with labour will be assessed using the Roberts coping with labour algorithm the midwife looks out for cues for coping and not coping
Length of labour | labour duration
  From time of admission (4-6cm) to birth
Apgar score | At 1 and 5 minutes
  Apgar score of baby at birth
use of oxytocin to augment labor | labor duration
  Use of oxytocin to augment labor
Maternal satisfaction questionnaire | Labour duration
  Level of satisfaction on support, information, pain control, humaneness and general satisfaction with birthing experience

CONTACTS AND LOCATIONS:
Overall Officials: Gorrette Nalwadda, PhD, Study Chair — Makerere University
Locations (1):
- Mbale Regional Referral Hospital, Mbale, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wanyenze EW, Nalwadda GK, Tumwesigye NM, Byamugisha JK. Efficacy of midwife-led role orientation of birth companions on maternal satisfaction and birth outcomes: a randomized control trial in Uganda. BMC Pregnancy Childbirth. 2023 Sep 18;23(1):669. doi: 10.1186/s12884-023-05978-8. PMID 37723430